CLINICAL TRIAL: NCT04638881
Title: A Prospective, Randomized, Double-blind, Placebo-controlled Trial of the Effects of Magnesium Sulfate on Postoperative Esophageal Spasm-associated Pain Following Peroral Endoscopic Myotomy
Brief Title: Magnesium for Peroral Endoscopic Myotomy
Acronym: MgPOEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Richard K. Kim, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58859
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Spasm
MeSH Terms: conditions — Esophageal Spasm, Diffuse | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Magnesium sulfate 50 mg/kg bolus + 25 mg/kg/hr infusion (Experimental): Bolus to be administered at start of mucosal incision, followed by infusion. Infusion to be terminated at extubation.
  Interventions: Drug: Magnesium sulfate
- Normal saline 0.9% 50 mg/kg bolus + 25 mg/kg/hr infusion (Placebo Comparator): Bolus to be administered at start of mucosal incision, followed by infusion. Infusion to be terminated at extubation.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Magnesium sulfate — Magnesium infusion 50 mg/kg bolus over 15 minutes and 25 mg/kg/hr infusion, both administered intraoperatively under general anesthesia.
  Arms: Magnesium sulfate 50 mg/kg bolus + 25 mg/kg/hr infusion
Drug: Normal Saline — Placebo. Bolus and infusion administered similarly under general anesthesia.
  Arms: Normal saline 0.9% 50 mg/kg bolus + 25 mg/kg/hr infusion

SUMMARY:
Postoperative pain after peroral endoscopic myotomy occurs due to involuntary esophageal smooth muscle spasms. Magnesium has antispasmodic properties as a smooth muscle relaxant. This study hypothesizes that among patients having peroral endoscopic myotomy, magnesium will decrease postoperative esophgeal pain as measured by the esophageal symptoms questionnaire, while decreasing perioperative opioid requirements.

ELIGIBILITY:
Inclusion Criteria:

- Planned peroral endoscopic myotomy procedure

Exclusion Criteria:

* cannot give consent
* patients who are clinically unstable and/or require urgent/emergent intervention
* previous esophageal myotomy
* preexisting hypermagnesemia
* end-stage renal disease
* neuromuscular disease, including but not limited to Guillain-Barre syndrome, myasthenia gravis, congenital myopathy, and muscular dystrophy
* preexisting heart failure
* severe ventricular systolic dysfunction (left or right ventricle)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Kim, MD, Principal Investigator — Stanford University; Joo H Hwang, MD PhD, Principal Investigator — Stanford University; Ban C Tsui, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnesium Sulfate 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Normal Saline 0.9% 50 mg/kg Bolus + 25 mg/kg/hr Infusion
Started | 46 | 46
Completed | 46 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Sulfate 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Normal Saline 0.9% 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (18) | 58 (18) | 58 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 19 | 19 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92
Body Mass Index (units: kg / m2) [Mean (Standard Deviation); unit: kg/m^2] | 25.6 (7.5) | 26.4 (7.0) | 26.1 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Esophageal Symptoms Questionnaire Score (ESQ)
Description: ESQ score is a validated survey score based on questions evaluating esophageal dysphagia, globus, and reflux. Participants answer 11 questions, each rated on a scale of 1 (Not severe) to 7 (Very severe). Scores were summed for an overall score (range 11 to 77, higher scores indicate more severe dysphagia).
Time Frame: 0 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Magnesium Sulfate 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Normal Saline 0.9% 50 mg/kg Bolus + 25 mg/kg/hr Infusion
Number analyzed (Participants) | 46 | 46
score on a scale | 24 [18 to 31] | 35 [28 to 42]

2. Secondary Outcome: Esophageal Symptoms Questionnaire Score (ESQ)
Description: as for outcome 1
Time Frame: 24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Magnesium Sulfate 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Normal Saline 0.9% 50 mg/kg Bolus + 25 mg/kg/hr Infusion
Number analyzed (Participants) | 46 | 46
score on a scale | 16 [14 to 23] | 30 [24 to 35]

3. Secondary Outcome: Postoperative Opioid Consumption
Description: Measured in oral morphine milliequivalents
Time Frame: From extubation to 24 hours after extubation
Measure: Median (Inter-Quartile Range); unit: morphine milliequivalents (MME)
Arm/Group | Magnesium Sulfate 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Normal Saline 0.9% 50 mg/kg Bolus + 25 mg/kg/hr Infusion
Number analyzed (Participants) | 46 | 46
morphine milliequivalents (MME) | 0 [0 to 4] | 30 [14 to 41]

4. Secondary Outcome: Postoperative Day 1 Opioid Consumption
Description: Measured in oral morphine milliequivalents
Time Frame: From 24 hours after extubation to 48 hours after extubation
Measure: Median (Inter-Quartile Range); unit: morphine milliequivalents (MME)
Arm/Group | Magnesium Sulfate 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Normal Saline 0.9% 50 mg/kg Bolus + 25 mg/kg/hr Infusion
Number analyzed (Participants) | 46 | 46
morphine milliequivalents (MME) | 0 [0 to 0] | 6 [0 to 20]

5. Secondary Outcome: Average Visual Acuity Score Pain Score in Postanesthesia Care Unit
Description: Pain measuring scale based on scale from 0 (no pain) to 10 (severe pain).
Time Frame: From extubation to discharge from postanesthesia care unit (up to 4 hours)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Magnesium Sulfate 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Normal Saline 0.9% 50 mg/kg Bolus + 25 mg/kg/hr Infusion
Number analyzed (Participants) | 46 | 46
score on a scale | 0 [0 to 3] | 5 [5 to 7]

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Magnesium Sulfate 50 mg/kg Bolus + 25 mg/kg/hr Infusion | Normal Saline 0.9% 50 mg/kg Bolus + 25 mg/kg/hr Infusion
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT04638881/Prot_SAP_000.pdf